CLINICAL TRIAL: NCT03560336
Title: Prospective, Multicentre, Open-label, Single-arm, Non-interventional Regulatory Post-marketing Surveillance(rPMS) Study to Evaluate the Safety and Effectiveness of Saxenda® (Liraglutide 3.0 mg) in Obese Patients and Overweight Patients With Obesity-related Comorbidities in Routine Clinical Practice in Korea
Brief Title: A Regulatory Post-marketing Surveillance (rPMS) Study to Evaluate the Safety and Effectiveness of Saxenda®(Liraglutide 3.0 mg) in Obese Patients and Overweight Patients With Obesity-related Comorbidities in Routine Clinical Practice in Korea.
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4380; U111-1199-8606 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall Population: Patients will be treated with commercially available liraglutide 3.0 mg according to routine clinical practice at the discretion of the treating physician
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Patients will initiate treatment with liraglutide according to the approved label in Korea. Patients will initiate 0.6 mg daily and weekly increase the dose by 0.6 mg until reaching 3.0 mg daily. Patients will then continue to stay on 3.0 mg/day (total treatment duration: 26 weeks).

SUMMARY:
The purpose of this study is to collect information about the safety and effectiveness of Saxenda® in obese patients and overweight patients with obesity-related comorbidities. The participant will attend the clinic or hospital according to usual practice and receive medical care, as agreed with the study doctor. The participation is expected to be approximately for 26 weeks.

ELIGIBILITY:
Inclusion Criteria: - The decision to initiate treatment with commercially available Saxenda® has been made by the patient/Legally Acceptable Representative (LAR) and the physician before and independently from the decision to include the patient in this study - Informed consent obtained before any study-related activities Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study - Male or Female of Native Korean, age greater than or equal to 18 years who is scheduled to start treatment with Saxenda® based on the clinical judgment of physician as specified in the Korean-Prescribing Information (local label) Exclusion Criteria: - Patients who are or have previously been on Saxenda® therapy - Known or suspected hypersensitivity to Saxenda® , the active substance or any of the excipients - Previous participation in this study. Participation is defined as having given informed consent in this study - Treatment with any investigational drug within 30 days prior to enrolment into the study - Female patient who is pregnant, breast-feeding, or intends to become pregnant and is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by Korea regulation or practice) - Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients and overweight patients with obesity-related comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 758 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) by preferred term (PT) | From baseline to week 13 (± 3 weeks)
  Count of events
Incidence of adverse events (AEs) by preferred term (PT) | From baseline to week 26 (± 3 weeks)
  Count of events

SECONDARY OUTCOMES:
Number of adverse drug reaction (ADRs) | From baseline to week 13 (± 3 weeks)
  Count of events
Number of adverse drug reaction (ADRs) | From baseline to week 26 (± 3 weeks)
  Count of events
Number of serious adverse events (SAEs) and serious adverse drug reations (SADRs) | From baseline to week 13 (± 3 weeks)
  Count of events
Number of serious adverse events (SAEs) and serious adverse drug reations (SADRs) | From baseline to week 26 (± 3 weeks)
  Count of events
Number of unexpected AEs and unexpected ADRs | From baseline to week 13 (± 3 weeks)
  Count of events
Number of unexpected AEs and unexpected ADRs | From baseline to week 26 (± 3 weeks)
  Count of events
Number of unexpected SAEs and unexpected SADRs | From baseline to week 13 (± 3 weeks)
  Count of events
Number of unexpected SAEs and unexpected SADRs | From baseline to week 26 (± 3 weeks)
  Count of events
Dose of liraglutide after administration initiation | week 13 (± 3 weeks)
  Measured in mg
Dose of liraglutide after administration initiation | week 26 (± 3 weeks)
  Measured in mg
Body weight loss (%) from week 0 to week 13 | Week 0, week 13
  Measured in percentage
Body weight loss (%) from week 0 to week 26 | Week 0, week 26
  Measured in percentage
Body weight loss (kg) from week 0 to week 13 | Week 0, week 13
  Measured in kg
Body weight loss (kg) from week 0 to week 26 | Week 0, week 26
  Measured in kg
The proportion of patients losing at least 5% of week 0 body weight at week 13 | Week 0, week 13
  Proportion of patients
The proportion of patients losing at least 5% of week 0 body weight at week 26 | Week 0, week 26
  Proportion of patients
The proportion of patients losing more than 10% of week 0 body weight at week 13 | Week 0, week 13
  Proportion of patients
The proportion of patients losing more than 10% of week 0 body weight at week 26 | Week 0, week 26
  Proportion of patients

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (11):
- South Korea (11):
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Gangwon-do
  - Novo Nordisk Investigational Site, Gwangju
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com